CLINICAL TRIAL: NCT01555216
Title: A Randomized Comparison of a Continuous Posterior Tibial Nerve Block and Single Injection Posterior Tibial Nerve Block in Patients Undergoing Forefoot Surgery
Brief Title: Continuous Tibial Nerve Block Versus Single Shot Tibial Nerve Block
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participant recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Associate Professor in Anesthesiology and Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00037311
Record Dates: First submitted 2011-10-20; First posted 2012-03-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Hallux Valgus
Keywords: Forefoot surgery
MeSH Terms: conditions — Hallux Valgus | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior tibial nerve catheter (Active Comparator): 5 ml bolus of 0.5% ropivacaine. The catheter will then be connected to a portable pump delivering 3 ml/h of 0.2% ropivacaine with a 2ml bolus every two hours.
  Interventions: Drug: Posterior tibial nerve catheter
- Single injection PTNB (Active Comparator): Single injection posterior tibial nerve block (PTNB) of 0.5% ropivacaine
  Interventions: Drug: Single injection posterior tibial nerve block

INTERVENTIONS:
Drug: Single injection posterior tibial nerve block — 5 ml of 0.5% ropivacaine
  Other Names: Naropin
  Arms: Single injection PTNB
Drug: Posterior tibial nerve catheter — 5ml bolus of 0.5% ropivacaine with 3 ml/h of 0.2% ropivacaine with a bolus every two hours
  Other Names: Naropin
  Arms: Posterior tibial nerve catheter

SUMMARY:
Foot surgery often causes severe and prolonged pain postoperatively. Prior methods of postoperative pain control included oral narcotics, single injection regional techniques and more recently continuous nerve catheters. Recent studies have demonstrated a benefit with continuous popliteal catheters when compared to single injection techniques in regards to postoperative pain control and patient satisfaction for foot surgeries.

Nerve blocks in the popliteal fossa involve both the common peroneal nerve and the tibial nerve. The innervation to the plantar surface of the forefoot involves the tibial nerve and does not involve the peroneal nerve. The purpose of this study is to compare the continuous posterior tibial nerve catheter with a single injection posterior tibial nerve block when used as part of a surgical ankle block for forefoot surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 to 65 years old) undergoing elective scheduled forefoot surgery (hallux valgus repair and metatarsal osteotomy).

Exclusion Criteria:

* Patient refusal to be included
* Presence of language barrier that prohibits proper communication with patient
* Under age of 18,
* Pregnancy
* History of allergy to local anesthetics or opioids
* Presence of a progressive neurological deficit
* Chronic opioid or drug abuse
* Diabetes
* Active infection in leg
* Unstable cardiovascular, renal or hepatic disease,
* Unwillingness to comply with follow up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | Up to five days
  Quality of recovery

SECONDARY OUTCOMES:
Pain control (pain score) | Up to 1 week
  pain control (pain score) between groups
Opioid consumption | Up to 1 week
  Opioid consumption
patient satisfaction | Up to 1 week
  patient satisfaction with pain control

CONTACTS AND LOCATIONS:
Overall Officials: Antoun Nader, MD, Principal Investigator — Northwestern Memorial Hospital
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No